CLINICAL TRIAL: NCT04680962
Title: A Double-Blind, Randomized, Parallel-Group Study to Investigate the Pharmacokinetic and Clinical Similarity Between MabionCD20, EU-approved MabThera® and US-licensed Rituxan® in Patients With Moderate-to-Severe Rheumatoid Arthritis
Brief Title: MabionCD20® Compared to MabThera® and Rituxan® in Patients With Rheumatoid Arthritis
Acronym: MABRIDGE
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study closed for business reasons before patient recruitment was initiated.
Sponsor: Mabion SA (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MabionCD20-003RA
Record Dates: First submitted 2020-12-02; First posted 2020-12-23 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Rituximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- MabionCD20 / MabionCD20 (Experimental): Patients receive one or two treatment courses of MabionCD20, each consisting of two 1000 mg i.v. infusions at an interval of 14 days. Investigational drug will be administered at Day 1 and Day 15, and, if patient is eligible for re-treatment, also at Week 24 and Week 26.
  Interventions: Biological: MabionCD20 (candidate biosimilar to rituximab)
- EU-Rituximab / EU-Rituximab (Active Comparator): Patients receive one or two treatment courses of MabThera®, each consisting of two 1000 mg i.v. infusions at an interval of 14 days. Investigational drug will be administered at Day 1 and Day 15, and, if patient is eligible for re-treatment, also at Week 24 and Week 26.
  Interventions: Biological: MabThera®
- US-Rituximab / MabionCD20 (Active Comparator): Patients receive a single treatment course of Rituxan®, consisting of two 1000 mg i.v. infusions at Day 1 and Day 15. After 24 weeks of follow-up, all patients eligible for re-treatment, are switched to receive a single treatment course of MabionCD20, consisting of two 1000 mg i.v. infusions at Week 24 and Week 26.
  Interventions: Biological: MabionCD20 (candidate biosimilar to rituximab); Biological: Rituxan®

INTERVENTIONS:
Biological: MabionCD20 (candidate biosimilar to rituximab) — Intravenous infusion, 10 mg/ml concentrate, 500 ml
  Other Names: Rituximab Mabion
  Arms: MabionCD20 / MabionCD20; US-Rituximab / MabionCD20
Biological: MabThera® — Intravenous infusion, 10 mg/ml concentrate, 500 ml
  Other Names: EU-Rituximab
  Arms: EU-Rituximab / EU-Rituximab
Biological: Rituxan® — Intravenous infusion, 10 mg/ml concentrate, 500 ml
  Other Names: US-Rituximab
  Arms: US-Rituximab / MabionCD20

SUMMARY:
Primary objective of the study is to establish a 3-way PK similarity bridge between MabionCD20 (candidate biosimilar to rituximab), MabThera® (EU-sourced rituximab) and Rituxan® (US-sourced rituximab) following the administration of these drugs to patients with moderate-to-severe rheumatoid arthritis. Main secondary objective is to confirm therapeutic similarity between MabionCD20 and the reference rituximab.

DETAILED DESCRIPTION:
Patients with active moderate-to-severe rheumatoid arthritis diagnosed according to the 2010 ACR criteria will be randomized to receive a blinded treatment course of either MabionCD20, EU-Rituximab (MabThera®) or US-Rituximab (Rituxan®) on the top of a stable methotrexate therapy. Two infusions of investigational drug at a dose of 1000 mg will be given at Day 1 and 15. Patients will be then followed for a minimum of 24 weeks to establish PK and therapeutic similarity and to compare PD, safety and immunogenicity parameters between the three rituximab products (Main Phase). Patients may receive a second course of investigational therapy at Week 24, provided that they meet re-treatment eligibility criteria specified in the study protocol. Subjects in MabionCD20 and EU-Rituximab groups will be continued on their assigned treatments, while all subjects in US-Rituximab group will be switched to MabionCD20. All subjects (re-treated and not re-treated) will continue the follow-up until Week 48 to collect long-term safety, immunogenicity and efficacy data.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Male or female, age 18 - 80 years
2. Body Surface Area (BSA) between 1.5 and 2.2 m2
3. Confirmed diagnosis of RA diagnosed according to the revised (2010) ACR/EULAR classification criteria, with a disease duration minimum of 6 months prior to the Screening Visit
4. Currently moderate to severe RA despite ongoing administration of an adequate MTX regimen. Moderate to severe disease is defined here as the presence of the following two criteria:

   1. Six or more swollen joints and ≥6 tender/painful joints, verified by a physician during the screening and re-confirmed at baseline visit (Day 1)
   2. DAS28 score ≥3.2 at screening
5. No history of treatment with TNF-α inhibitor (innovative or biosimilar, authorized or investigational) at any time before the screening i.e. TNF-α inhibitor naive population.
6. Receiving MTX treatment at a dosage of 7.5-25 mg/week for at least 12 weeks prior to screening, with the last 4 weeks at a stable dose, and willing to remain at this dose for the entire study duration
7. Male or WOCBP must consent to use highly effective contraception, from the Screening Visit, during the intervention period, and for at least 12 months after the last dose of study intervention
8. Female participants must not be pregnant or lactating (negative baseline serum test)

EXCLUSION CRITERIA:

1. History of or current inflammatory joint disease other than RA
2. History of or current systemic autoimmune disorder
3. ACR functional class IV disease
4. History of psychiatric disorder that would interfere with normal participation in the study
5. Evidence of HBV, HCV, HIV infection
6. Evidence of laboratory-confirmed or clinically suspected SARS-CoV-2 infection within 14 days before the study drug administration and a documented positive RT-PCR test within 72 hours before the first infusion or positive antigen test within 24 hours before the first infusion.
7. Serious and/or uncontrolled coexisting diseases which are recognized as major contraindications to the administration of rituximab, methotrexate or any of the pre-medication components or as important risk factors for the development of severe or life-threatening SARS-CoV-2 infection or other factors, which in the Investigator's opinion, would preclude patients participation. This category includes severe pulmonary, cardiovascular, neurologic, renal and hepatic diseases, severe and inadequately controlled type 1 or 2 diabetes.
8. Recent history or current evidence of bacterial, viral or fungal infection (excluding infections of nailbeds)
9. History of or current active tuberculosis, with typical symptoms of M. tuberculosis infection confirmed by positive results of TB screening test or documented diagnosis prior to screening
10. Latent tuberculosis, as documented in subject's medical records or shown by a positive or indeterminate QuantiFERON test performed at screening, in absence of typical symptoms of tuberculosis. However, a patient with latent tuberculosis may become eligible for the study if he/she meets the following criteria:

    1. Patient completed a standard TB prophylaxis prior to the screening and had no active TB or contact with active TB case after completion of the most recent prophylactic regimen OR received at least four weeks of standard TB prophylactic regimen prior to the screening visit and is capable and willing to continue on this regimen while participating in the study.
    2. Patient has no active TB at the time of screening, which must be confirmed through referral to a TB specialist if > 1 year has passed since the completion of the last prophylaxis or if the prophylaxis is still being received by the time of screening
    3. Patient had no positive findings on chest X-ray examination at screening and within three months prior to screening
11. History of cancer (solid tumors, hematologic malignancies and other) within 5 years of the screening
12. History of significant cytopenia or other disorder of the hematopoietic system
13. Primary or secondary immunodeficiency
14. Any other condition that is listed as a contraindication to receive rituximab or methotrexate therapy
15. Recent use of biologic DMARDs or non-biologic DMARDs other than MTX within the washout periods specified in the study protocol
16. Treatment with any of the authorized or investigational TNF-α inhibitors at any time before the screening (regardless if innovative or biosimilar).
17. History of prior treatment with a B cell modulating or B cell depleting therapy such as, but not limited to, rituximab or other anti CD20 mAb (ocrelizumab, ofatumumab, obinutuzumab), belimumab, atacicept, tabalumab, epratuzumab and other experimental treatments
18. Use of systemic glucocorticoids at a dose higher than 10 mg prednisolone daily or equivalent, within 2 weeks prior to Screening or between screening and Day 1
19. Use of intraarticular hyaluronic acid injection within 28 days before the screening or between screening and Day 1.
20. Use of any drug that has not received regulatory approval for any indication within 4 weeks or a minimum of 5 half-lives, whichever is longer, prior to the Screening Visit or planned receipt of unauthorized drug or vaccine during the study.
21. History of prior allergic or anaphylactic reaction to rituximab therapy (or to any excipient contained in the study IMP)
22. Serious abnormal laboratory findings, specifically:

    1. White blood cell count <3,000/μL OR neutrophil count <1,500/μL.
    2. Platelet count <75,000/μL.
    3. Aspartate aminotransferase or alanine aminotransferase >2.5 times ULN.
    4. Hemoglobin <8.0 g/dL.
    5. IgG below 5.0 mg/mL or IgM below 0.4 mg/mL.
    6. Any other clinically significant laboratory abnormality.
23. Intolerance or contraindications to administration of MTX therapy, i.v. glucocorticoids, or to any other component of the premedication
24. Major surgery (including joint surgery) within 8 weeks prior to Screening or planned surgery within 12 months after baseline
25. Recent vaccination with inactivated/non-live vaccine (<4 weeks prior to study intervention infusion on Day 1) or live vaccine (<6 weeks prior to study intervention infusion on Day 1) vaccine
26. Planned vaccination with live vaccine during the follow-up.
27. Chronic intake of narcotic analgesics (e.g. morphine, fentanyl, hydrocodone, oxycodone, codeine).
28. Participation in a clinical study during the 2 months prior to enrolment in the study (exemption - previously failed screening procedures in MabionCD20-003RA study).
29. Female patients breastfeeding, pregnant or planning of pregnancy within 12 months after the last infusion of the study intervention.
30. Blood donation or other blook loss of more than 500 ml within the last two months prior to Screening Visit.
31. Lack of peripheral venous access.
32. History of drug, alcohol or chemical abuse within 2 years prior to screening.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-08-03 (Actual); Primary Completion 2023-08-03 (Actual); Study Completion 2023-08-03 (Actual)

PRIMARY OUTCOMES:
Area Under the Serum Concentration-time Curve from Day 1 to Week 24, with extrapolation to infinity [AUC 0-inf (D1-W24)] | Day 1 to Week 24
  Concentration of rituximab in serum over the entire PK study duration, with extrapolation to infinity. Outcome based on all PK samples collected in the study - from Day 1 (first infusion) to Week 24 (before administration of the 2nd treatment course).
Area Under the Serum Concentration-time Curve from Day 1 to Day 15 [AUC 0-t (D1-D15)] | Day 1 to Day 15
  Concentration of rituximab in serum measured from Day 1 (before the 1st drug infusion) to Day 15 (before the 2nd drug infusion).

SECONDARY OUTCOMES:
Mean Change from Baseline in DAS28-ESR score | Baseline to Week 48
  DAS28-ESR is a disease activity index calculated from the following variables:
  * Tender joint count (28 joints);
  * Swollen joint count (28 joints);
  * Erythrocyte sedimentation rate (ESR);
  * Patient's assessment of global disease activity.
  The score ranges from 0 to ca. 10 points, with > 5.1 indicating high disease activity, < 3.2 indicating low disease activity, and < 2.6 indicating clinical remission. Change from baseline to Week 24 will be used for the confirmation of therapeutic similarity.
  For the US submission, therapeutic similarity will be confirmed if 90% CI of the difference between MabionCD20 and the combined EU- plus US-Rituximab group is contained within (-0.6; +0.5) equivalence margin. For the EU submission, therapeutic similarity will be declared if 95% CI of the difference is contained within (-0.6; +0.6) margin. In an additional analysis, MabionCD20 group will be compared against EU-Rituximab group alone using the above EU criteria.
Mean Change from Baseline in DAS28-CRP score | Baseline to Week 48
  DAS28-CRP is a disease activity index calculated from the following variables:
  * Tender joint count (28 joints);
  * Swollen joint count (28 joints);
  * C-reactive protein (CRP);
  * Patient's assessment of global disease activity.
  It ranges from 0 to ca. 10 points, with a score > 5.1 indicating high disease activity, a score < 3.2 indicating low disease activity, and a score < 2.6 indicating clinical remission of RA.
Percentage of patients achieving an ACR20/50/70 response | Baseline to Week 48
  A positive ACR20/50/70 response is achieved, when all of the following improvement criteria are met:
  1. ≥ 20%/50%/70%* improvement in tender joint count.
  2. ≥ 20%/50%/70%* improvement in swollen joint count.
  3. ≥ 20%/50%/70%* improvement in minimum 3 of the following 5 parameters:
     * Patient's assessment of pain;
     * Patient's global assessment of disease activity;
     * Physician's global assessment of disease activity;
     * Patient's assessment of physical function (HAQ-DI);
     * Laboratory evaluation of acute phase reactant (ESR)
       * 20%, 50% and 70% improvement apply to ACR20, ACR50 and ACR70 response, respectively
Percentage of patients with low disease activity (DAS28-ESR <3.2) | Baseline to Week 48
  DAS28 scale ranges from 0 to approximately 10 points, with a score higher than 5.1 indicating high disease activity, a score less than 3.2 indicating low disease activity, and a score less than 2.6 indicating clinical remission of RA.
Percentage of patients with disease remission (DAS28-ESR <2.6) | Baseline to Week 48
  DAS28 scale ranges from 0 to approximately 10 points, with a score higher than 5.1 indicating high disease activity, a score less than 3.2 indicating low disease activity, and a score less than 2.6 indicating clinical remission of RA.
Percentage of patients with a moderate response on EULAR scale | Baseline to Week 48
  There are three categories of EULAR response (good, moderate and non-responders) which include not only the individual's amount of change in the DAS but also the attainment of a particular DAS value (low, moderate or high) at the endpoint.
  To be classified as having a moderate EULAR response, the patient must demonstrate a minimum change from baseline on DAS28-ESR of > 0.6 to < 1.2, as well as the endpoint achievement of a DAS-28 ≤ 5.1.
Percentage of patients with a good response on EULAR scale | Baseline to Week 48
  There are three categories of EULAR response (good, moderate and non-responders) which include not only the individual's amount of change in the DAS but also the attainment of a particular DAS value (low, moderate or high) at the endpoint.
  To be classified as having a good EULAR response, the patient must demonstrate a significant change from baseline (> 1.2) as well as reach low disease activity (DAS-28 ≤ 3.2).
Simplified Disease Activity Index (SDAI) | Baseline to Week 48
  SDAI is composed of the following clinical and laboratory variables:
  * tender joint count (up to 28 joints);
  * swollen joint count (up to 28 joints);
  * patient's assessment of global disease activity;
  * physician's assessment of global disease activity;
  * CRP (C-reactive protein).
  Summation of all above variables produces a SDAI score (maximum 86.0 points). High disease activity is defined on SDAI as a score higher than 26.0 points, while a cut-off for remission is set at 3.3 points.
Clinical Disease Activity Index (CDAI) | Baseline to Week 48
  CDAI is calculated in the same way as SDAI, except that only clinical parameters of disease level are taken into account (without CRP). Maximum score is 76.0 points. High disease activity is defined above 22.0 points and remission as ≤ 2.8 points
Area Under the Serum Concentration-time Curve from Day 1 to Week 24 [AUC 0-t (D1-W24)] | Baseline to Week 24
  Concentration of rituximab in serum over the entire PK study duration, without extrapolation to infinity. Outcome based on all PK samples collected in the study - from Day 1 (first infusion) to Week 24 (before administration of the 2nd treatment course).
Area Under the Serum Concentration-time Curve from Day 15 to Week 24 [AUC 0-t (D15-W24)] | Day 15 to Week 24
  Concentration of rituximab in serum measured from Day 15 (before the 2nd drug infusion) to Week 24 (before the 2nd treatment course)
Maximum drug concentration in serum after the 1st infusion (Cmax1) | Day 1
  Maximum drug concentration measured after the 1st study drug infusion at Day 1
Maximum drug concentration in serum after the 2nd infusion (Cmax2) | Day 15
  Maximum drug concentration measured after the 2nd study drug infusion at Day 15
Trough drug concentration in serum (Ctrough) | Day 15
  Drug concentration measured shortly before the 2nd study drug infusion at Day 15
Time to achieve maximum drug concentration in serum after the 1st infusion (Tmax1) | Day 1
  Time to achieve maximum drug concentration in serum after the 1st infusion at Day 1
Time to achieve maximum drug concentration in serum after the 2nd infusion (Tmax2) | Day 15
  Time to achieve maximum drug concentration in serum after the 2nd infusion at Day 15
Absolute CD19+ B cell counts by visit | Day 1 to Week 24
  Evolution of CD19+ B cell counts from the 1st study drug infusion at Day 1 to Week 24
Percentage of patients with undetectable levels of CD19+ B-cells | Day 3 and Week 24
  Percentage of patients who achieve a complete depletion of CD19+ B-cells two days after the 1st infusion (Day 3) and percentage of patients who remain depleted of CD19+ B-cells on Week 24
Percentage of patients with Adverse Events (AEs) | Day 1 to Week 48
  Patients with AEs, which occurred after signing the Informed Consent Form (ICF) until the study end at Week 48. Several categories of AEs will be evaluated:
  * Treatment-emergent adverse events (TEAEs, AEs occurring after the initiation of study treatment);
  * Related TEAEs (classified as at least possibly related to the study drug by Investigators);
  * Severe TEAEs;
  * TEAEs leading to permanent/temporary discontinuation of the study drug or reduction in infusion rate;
  * Treatment-emergent serious adverse events (TESAEs);
  * Related TESAEs;
  * TESAEs leading to permanent/temporary discontinuation or reduction in infusion rate;
  * TEAEs leading to death;
  * Adverse events of special interest (AESI), which include: Infusion-related reactions (IRRs), Hypersensitivity and allergic reactions, Infusion-associated cardiovascular events, Serious infection events, SARS-CoV-2 infections and Progressive multifocal leukoencephalopathy (PML).
Percentage of patients with a positive anti-drug antibody (ADA) response | Day 1 to Week 48
  Positive ADA response is a composite of treatment-induced and treatment-boosted ADAs. Patients with persistent response will be distinguished from patients with transient ADAs. Patients with positive samples will be additionally analyzed for ADA titer and for the presence of drug neutralizing antibodies (percentage of patients with nAb).

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Sponsor's website — https://www.mabion.eu